CLINICAL TRIAL: NCT00590447
Title: Treatment of Patients With Posttransplant Lymphoproliferative Disorder (PTLD) With a Sequential Treatment Consisting of Anti-CD20 Antibody Rituximab and CHOP+GCSF Chemotherapy (PTLD-1/3)
Brief Title: Risk Stratified Sequential Treatment for CD20-positive PTLD
Acronym: PTLD-1/3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Ralf Trappe, Head German PTLD Study Group, Charite University, Berlin, Germany
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PTLD-1, 3rd. amendment; EudraCT 2005-000743-29
Record Dates: First submitted 2007-12-28; First posted 2008-01-10 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2017-03

CONDITIONS: PTLD; Posttransplant Lymphoproliferative Disorder
Keywords: 1st-line therapy; single agent rituximab; CHOP; risk stratification

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): All patients will receive 4 courses of rituximab on days 1, 8, 15 and 22. Patients achieving a CR after the first 4 applications of single agent rituximab (evaluated between day 40 to 50) will go on with 4 further courses of single agent rituximab on days 50, 72, 94 and 116.
  Interventions: Drug: rituximab monotherapy
- B (Experimental): All patients will receive 4 courses of rituximab on days 1, 8, 15 and 22. Patients who do not achieve a CR after the first 4 applications of single agent rituximab (evaluated between day 40 to 50) will go on with 4 courses of R-CHOP on days 50, 72, 94 and 116.
  Interventions: Drug: sequential R-CHOP

INTERVENTIONS:
Drug: rituximab monotherapy — 375 mg/m2, IV on days 1, 8, 15, 22, 50, 72, 94 and 116. In case of disease progression during the first 4 administration of rituximab antibody or the 4 weeks interval between course 4 and 5 the patients directly enter R-CHOP chemotherapy (Arm B).
  Arms: A
Drug: sequential R-CHOP — 375 mg/m2 rituximab, IV on days 1, 8, 15, 22, 50, 72, 94 and 116. Cyclophosphamid 750 mg/m2, adriamycine 50 mg/m2 and vincristine 1.4mg/m2, IV and prednisone 50mg/m2, PO every 3 weeks at days 50, 72, 94 and 116.
  In case of disease progression during the first 4 administration of rituximab antibody or the 4 weeks interval between antibody and R-CHOP administration the patients directly enter R-CHOP chemotherapy.
  Arms: B

SUMMARY:
This phase-II trial will investigate the efficacy, safety and the tolerability of a sequential therapy consisting of 4 courses of single agent rituximab followed by 4 courses of R-CHOP chemotherapy in patients with CD20+ posttransplant lymphoproliferative disorders (PTLD). However, responders to rituximab achieving a CR after the first 4 applications of rituximab will go on with rituximab monotherapy and will not receive chemotherapy.

DETAILED DESCRIPTION:
The rationale for performing the present study is to combine two highly active treatment modalities in first line therapy of solid organ recipients with B-cell PTLD. The monoclonal antibody CD20 represents an effective therapeutic approach in the treatment of PTLD. Unfortunately this effect seems to be of limited duration in some patients, who benefited from monotherapy with rituximab. The advantage of this therapeutic approach in PTLD is due to the low incidence of third to fourth degree adverse events. At diagnosis of PTLD a relevant proportion of these patients is not suitable for first line cytotoxic chemotherapy due to widespread disease, organ dysfunction or reduced performance state. Insufficiencies of kidney or bone marrow function are frequent in organ recipients due the toxic side effects of the immunosuppressive drugs. After pre-phase treatment with the monoclonal antibody rituximab the CHOP chemotherapy is suggested to be less toxic due to the lower tumor burden. Thereby treatment related severe or even lethal toxicities, frequently reported in patients with PTLD who underwent cytotoxic chemotherapy, may be prevented. Furthermore the total number of cytotoxic cycles of CHOP-therapy is reduced from 6 for 8 to 4 cycles and thus may result in an additional reduction of toxicity in the single patient. Because immunochemotherapy (R-CHOP) is clearly superior to CHOP with respect to progression free survival and relapse rates in patients with classical NHL and rituximab is very unlikely to add any further toxicity to CHOP the majority of patients will go on with four courses of R-CHOP. However, patients with a complete remission after 4 courses of single agent rituximab may have a very favourable risk profile and therefore will go on with rituximab single agent instead of R-CHOP.

ELIGIBILITY:
Inclusion Criteria:

* PTLD with or without EBV association, confirmed after biopsy or resection of tumor
* Measurable disease of > 2 cm in diameter and/or bone marrow involvement
* Patients having undergone heart, lung, liver, kidney, pancreas, small intestine transplantation or other or a combination of the organ transplantations mentioned
* Karnofsky scale >50% or ECOG ≤ 3
* Reduction of immunosuppression with or without antiviral therapy
* A complete surgical extirpation of tumor was not performed
* A radiation therapy was not performed
* Effective contraception for women in childbearing age
* Patient's written informed consent and written consent for data collection
* Patients are > 18 years (or ≥ 15 years with parental agreement )

Exclusion Criteria:

* Life expectancy less than 6 weeks
* Karnofsky-scale <50% or ECOG ≥ 3
* Treatment with rituximab before
* Known allergic reactions against foreign proteins
* Concomitant diseases, which exclude the administration of therapy as outlined by the study protocol
* non-compensated heart failure
* Dilatative cardiomyopathy
* Myocardial infarction during the last 6 months
* Severe non-compensated hypertension
* Severe non-compensated diabetes mellitus
* Renal insufficiency (creatinine more than 3-fold of the upper normal value), not related to lymphoma
* Hepatic insufficiency with transaminase values greater than 3-fold of the normal values and/or bilirubin levels >3.0 mg/dl, not related to lymphoma
* Clinical signs of cerebral dysfunction
* Women during the lactation period, pregnant or of childbearing potential not using a reliable contraceptive method
* Involvement of the central nervous system by the disease
* Severe psychiatric disease
* Known to be HIV positive
* Missing written informed consent of the patient

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2006-12; Primary Completion 2014-12 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
The primary objective is the evaluation of the efficacy.For this aim the overall objective response rates after therapy = complete and partial response and the duration of the response will be measured. | evaluated 4 weeks after comleting therapy

SECONDARY OUTCOMES:
The secondary objective is to determine the adverse events and tolerability of rituximab and/or chemotherapy. Furthermore, the long-term safety will be determined, especially the frequency of complicating infections and the overall survival. | within 2 years of follow up

CONTACTS AND LOCATIONS:
Overall Officials: Hanno Riess, MD, Principal Investigator — Charité, Campus Virchow-Klinikum Berlin, Germany; Ralf U Trappe, MD, Study Chair — Charité, Campus Virchow-Klinkum, Berlin, Germany
Locations (7):
- Princess Alexandra Hospital, Ipswich Rd, Woolloongabba, Qld 4102, Brisbane, Australia
- Catholic University of Leuven, Department of Hematology, Leuven, Belgium
- Hôpital Pitié-Salpétrière, Department of Hematology, 47-83 Boulevard de l'Hopital, Paris, France
- Charité - Universitätsmedizin Berlin, Campus Virchow Klinikum, Department of Hematology and Oncology, Augustenburger Platz 1, Berlin, Germany
- Div. Universitaria Ematologia e Terapie Cellulari, University of Torino, Torino, Italy
- Zakład Propedeutyki Onkologii, Gdańskiego Uniwersytetu Medycznego, Gdynia, Poland
- Sahlgrens hospital, Department of Hematology, Gothenburg, Sweden

REFERENCES:
- [Result] Trappe RU, Dierickx D, Zimmermann H, Morschhauser F, Mollee P, Zaucha JM, Dreyling MH, Duhrsen U, Reinke P, Verhoef G, Subklewe M, Huttmann A, Tousseyn T, Salles G, Kliem V, Hauser IA, Tarella C, Van Den Neste E, Gheysens O, Anagnostopoulos I, Leblond V, Riess H, Choquet S. Response to Rituximab Induction Is a Predictive Marker in B-Cell Post-Transplant Lymphoproliferative Disorder and Allows Successful Stratification Into Rituximab or R-CHOP Consolidation in an International, Prospective, Multicenter Phase II Trial. J Clin Oncol. 2017 Feb 10;35(5):536-543. doi: 10.1200/JCO.2016.69.3564. Epub 2016 Dec 19. PMID 27992268